CLINICAL TRIAL: NCT07180901
Title: Proactive Risk-based Optimization & Notifications for Treatment & Outcomes (PRONTO) in Head & Neck Cancer: A Strategy to Reduce Delays From Surgery to Post-Operative Adjuvant Therapy in Head and Neck Cancer
Brief Title: Proactive Risk-based Optimization & Notifications for Treatment & Outcomes in Head & Neck Cancer
Acronym: PRONTO-HN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Health Services Research
Other Study IDs: DSP-21047
Record Dates: First submitted 2025-08-04; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Oral Cancer , Oral Squamous Cell Carcinoma, Oral Cavity Cancer; Head &Amp;Amp; Neck Squamous Cell Carcinoma; Larynx Squamous Cell Carcinoma
Keywords: Surgery to post-operative radiation therapy interval; Treatment delays; Oral cavity cancer
MeSH Terms: conditions — Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Therapeutics; Treatment Outcome; RID

STUDY DESIGN:
Intervention Model Description: A quasi-experimental, interrupted time-series. Group A will be pre-intervention and group B is post-intervention.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (No Intervention): Pre-implementation of care coordination system.
- Group B (Experimental): Post-implementation of PRONTO-HN system:
  1. Pre-operative risk stratification of requiring adjuvant therapy using our predictive model, applied at tumor board. Patients stratified as fast-track vs normal-track.
  2. High-risk patients receive intensive preoperative and postoperative coordination. Low-risk patients are monitored but escalated rapidly if adverse pathology is detected. This includes:
     * pre-operative dental consultation for fast-track
     * pre-operative oncology consultation for fast-track with high-risk features
     * target pathology results 14 days post-operatively for fast-track
  3. Automated reminders and target dates sent to members of the multidisciplinary team.
  Interventions: Other: Proactive Risk-Based Optimization and Notifications for Treatment and Outcomes (PRONTO)

INTERVENTIONS:
Other: Proactive Risk-Based Optimization and Notifications for Treatment and Outcomes (PRONTO) — Post-implementation of PRONTO-HN system: 1. Pre-operative risk stratification of requiring adjuvant therapy using our predictive model, applied at tumor board. Patients stratified as fast-track vs normal-track. 2. High-risk patients receive intensive preoperative and postoperative coordination. Low-risk patients are monitored but escalated rapidly if adverse pathology is detected. This includes: - pre-operative dental consultation for fast-track - pre-operative oncology consultation for fast-track with high-risk features - target pathology results 14 days post-operatively for fast-track 3. Automated reminders and target dates sent to members of the multidisciplinary team.
  Arms: Group B

SUMMARY:
Delays between surgery and the initiation of post-operative radiotherapy (S-PORT) in head and neck cancer (HNC) patients are prevalent and associated with worse oncologic outcomes. This pilot study evaluates whether a proactive, automated care coordination system (PRONTO-HN) can improve adherence to recommended S-PORT intervals of ≤42 days at the Centre hospitalier de l'Université de Montréal (CHUM).

The study is a single-center, quasi-experimental, interrupted time-series design with two phases. Group A (control) includes patients treated before the intervention (using a prospectively maintained database from August 2024 to August 2025). Group B (intervention) includes patients treated with the new coordination system from September 2025 to September 2026.

The intervention includes automated alerts, multidisciplinary task coordination, and risk stratification based on a predictive model developed and published by our team. This model uses only pre-operative data to estimate the likelihood that a patient will require adjuvant therapy after surgery, stratifying patients into high- and low-risk categories. High-risk patients receive intensified coordination protocols, including early oncology and dental consultations and shorter target times for pathology results.

Primary objective: Reduce the proportion of patients with S-PORT > 42 days. Secondary/tertiary objectives: Reduce mean S-PORT time. Evaluate impacts on overall, locoregional, and disease-free survival in a 2- and 3-year follow up study.

Patients are identified at the time the operating room request is submitted. Demographic, clinical, and oncologic data are collected and stored securely in REDCap. As the intervention is administrative in nature and does not modify patient care, consent is waived.

Statistical analysis will evaluate the intervention's effect and identify predictors of delays. A sample of 38 patients per group provides adequate power to detect a drop in S-PORT > 42 days from 80% to 50%.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age 18 or older).
* Pathologically confirmed oral cavity or laryngeal squamous cell carcinoma.
* Diagnosed from July 2024 to September 2026.
* With planned primary intention surgical resection.
* With or without adjuvant therapy.
* Treated at the Centre Hospitalier de l'Université de Montréal.

Exclusion Criteria:

* Patients who do not end up receiving surgery.
* S-PORT > 180 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-10-21 (Estimated); Study Completion 2029-10-21 (Estimated)

PRIMARY OUTCOMES:
Surgery to post-operative radiotherapy time (S-PORT) | Day 1 of radiotherapy (assessed up to 12 weeks post-operatively)
  Number of days between surgery and start of radiotherapy (adjuvant)

SECONDARY OUTCOMES:
Overall survival | From date of surgery until the date of date from any cause (assessed up to 60 months)
  Event: Death (of any cause) Censor: Alive at last follow-up
Locoregional Survival | From date of surgery until the date of locoregional recurrence or death, whichever came first (assessed up to 60 months)
  Event: Locoregional recurrence (primary site or cervical node) or death Censored: Alive and without locoregional recurrence at last follow-up
Distant metastasis-free survival | The time from surgery to event. From date of surgery until the date of distant metastasis or death, whichever came first (assessed up to 60 months)
  Event: Distant metastasis or death Censored: Alive and without distant metastasis at last follow-up
Recurrence-Free Survival | From date of surgery until the date of locoregional recurrence or distant metastasis, whichever came first (assessed up to 60 months)
  Event: Any recurrence (local, regional, or distant) Censored: Recurrence-free at last follow-up. Death without recurrence also censored.
Disease-Free Survival | From date of surgery until the date of locoregional recurrence or distant metastasis or death, whichever came first (assessed up to 60 months)
  Event: Recurrence (any site) or death Censored: Alive and disease-free at last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Houda Bahig, MD PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dayan GS, Bahig H, Colivas J, Eskander A, Johnson-Obaseki S, Chandarana S, de Almeida JR, Nichols AC, Hier M, Belzile M, Avagnina A, Hong X, Gaudet M, Matthews TW, Hart R, Goldstein DP, Hosni A, MacNeil D, Fowler J, Khalil C, Khoury M, Morand G, Sultanem K, Ayad T, Christopoulos A. Preoperative Clinical and Tumor Factors Associated With Adjuvant Therapy for Oral Cavity Cancer. JAMA Otolaryngol Head Neck Surg. 2025 May 1;151(5):466-475. doi: 10.1001/jamaoto.2024.5250. PMID 40146171
- [Background] Dayan G, Bahig H, Fortin B, Filion E, Nguyen-Tan PF, O'Sullivan B, Charpentier D, Soulieres D, Gologan O, Nelson K, Letourneau L, Schmittbuhl M, Ayad T, Bissada E, Guertin L, Tabet P, Christopoulos A. Predictors of prolonged treatment time intervals in oral cavity cancer. Oral Oncol. 2023 Dec;147:106622. doi: 10.1016/j.oraloncology.2023.106622. Epub 2023 Nov 8. PMID 37948896
- [Background] Dayan GS, Bahig H, Johnson-Obaseki S, Eskander A, Hong X, Chandarana S, de Almeida JR, Nichols AC, Hier M, Belzile M, Gaudet M, Dort J, Matthews TW, Hart R, Goldstein DP, Yao CMKL, Hosni A, MacNeil D, Fowler J, Higgins K, Khalil C, Khoury M, Mlynarek AM, Morand G, Sultanem K, Maniakas A, Ayad T, Christopoulos A. Oncologic Significance of Therapeutic Delays in Patients With Oral Cavity Cancer. JAMA Otolaryngol Head Neck Surg. 2023 Nov 1;149(11):961-969. doi: 10.1001/jamaoto.2023.1936. PMID 37422839

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT07180901/Prot_SAP_000.pdf